CLINICAL TRIAL: NCT06475716
Title: Efficacy of a Guided Internet-based Trauma-focused CBT Intervention 'Spring' for ICD-11 Posttraumatic Stress Disorder Symptoms: A Randomized Controlled Trial
Brief Title: Guided Internet-based Trauma-focused CBT Programme for Post-traumatic Stress Disorder 'Spring'
Acronym: SPRING-LT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vilnius University (Other)
Collaborators: Cardiff University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S-MIP-23-14
Record Dates: First submitted 2024-06-17; First posted 2024-06-26 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Posttraumatic Stress Disorder
Keywords: trauma; posttraumatic stress; treatment; cognitive behavior therapy; internet-based intervention
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to the immediate treatment group or delayed treatment control group. The immediate treatment group will receive the intervention immediately after randomization. The delayed treatment group will receive the intervention 22 weeks after randomization.
Who Masked: Outcomes Assessor
Masking Description: Semi-structured interviews will be administered by researchers blind to randomization allocation at baseline, 10 and 22 weeks after randomization. Self-report data will be collected via a secure online platform, so it will help avoid ascertainment bias in the measurement of outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate treatment group (Experimental): The immediate treatment group will receive the intervention immediately after randomization. The intervention includes using an online guided self-help programme Spring that is based on the principles of trauma-focused cognitive behavioral therapy and consists of 8 steps. The user of the programme also receives up to 3 hours of guidance by a trained therapist.
  Interventions: Behavioral: Internet-based guided programme Spring
- Delayed treatment control group (Active Comparator): The delayed treatment group will receive the same intervention as the immediate treatment group, but 24 weeks after randomization. The intervention includes using an online guided self-help programme Spring that is based on the principles of trauma-focused cognitive behavioral therapy and consists of 8 steps. The user of the programme also receives up to 3 hours of guidance by a trained therapist.
  Interventions: Behavioral: Internet-based guided programme Spring

INTERVENTIONS:
Behavioral: Internet-based guided programme Spring — Spring is an online guided self-help programme based on the principles of trauma-focused cognitive behavioral therapy and consists of 8 steps designed for delivery over 8 weeks. The steps cover psychoeducation, grounding techniques, management of anxiety, behavioral activation, imaginal exposure, cognitive restructuring, in vivo exposure, and prevention of relapse. The user of the programme also receives up to 3 hours of therapist guidance.

SUMMARY:
The main aim of the study is to evaluate the efficacy of the Lithuanian version of the internet-based guided self-help programme (Spring) in reducing ICD-11 PTSD symptoms.

DETAILED DESCRIPTION:
Spring is an online guided self-help programme for the reduction of posttraumatic stress disorder symptoms. It is based on the principles of trauma-focused cognitive behavioral therapy and consists of 8 steps covering psychoeducation, grounding techniques, management of anxiety, behavioral activation, imaginal exposure, cognitive restructuring, in vivo exposure, and prevention of relapse. The user of the programme also receives up to 3 hours of therapist guidance. Originally Spring was developed by the research team at Cardiff University. In the current study, the most recent second version of the Spring programme adapted to the Lithuanian population will be used. The main aim of the study is to evaluate the efficacy of the Lithuanian version of the Spring programme in reducing ICD-11 posttraumatic stress disorder symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or over
* Ability to read and write fluently in Lithuanian
* Have regular access to a device with an internet connection to use the programme
* Provide informed consent for participation
* Experience PTSD symptoms followed by a non-prolonged and non-repetitive traumatic experience as measured by the ITI

Exclusion Criteria:

* Regularly seeing a therapist or counsellor for mental health issues
* Change in psychotropic medication in the last month
* CPTSD diagnosis
* Psychosis
* Severe suicide risk
* Substance dependence
* Experiencing ongoing threat

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-09-10 (Estimated); Primary Completion 2025-12-20 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
Change in International Trauma Interview (ITI) PTSD score post-treatment | baseline; 10 weeks after randomization
  The ITI is a semi-structured clinical interview for the assessment of symptoms of ICD-11 posttraumatic stress disorder. The total ITI score measuring symptoms of PTSD may range from 0 to 24. Higher scores indicate greater symptom severity.

SECONDARY OUTCOMES:
Change in International Trauma Interview (ITI) PTSD score at a three-month follow-up | baseline; 22 weeks after randomization
  The ITI is a semi-structured clinical interview for the assessment of symptoms of ICD-11 posttraumatic stress disorder and disturbances is self organization (DSO). The total ITI score measuring DSO symptoms may range from 0 to 24. Higher scores indicate greater symptom severity.
Change in International Trauma Interview (ITI) DSO score | baseline; 10 weeks after randomization; 22 weeks after randomization
  The ITI is a semi-structured clinical interview for the assessment of symptoms of ICD-11 posttraumatic stress disorder and disturbances is self organization (DSO). The total ITI score measuring DSO symptoms may range from 0 to 24. Higher scores indicate greater symptom severity.
Change in International Trauma Questionnaire (ITQ) score | baseline; 10 weeks after randomization; 22 weeks after randomization; 32 weeks after randomization (delayed treatment group only)
  The ITQ is a self-report questionnaire for the assessment of symptoms of ICD-11 posttraumatic stress disorder and complex posttraumatic stress disorder. The overall ITQ score ranges from 0 to 24. Higher scores indicate greater symptom severity.
Change in International Depression Questionnaire (IDQ) score | baseline; 10 weeks after randomization; 22 weeks after randomization; 32 weeks after randomization (delayed treatment group only)
  The IDQ is a self-report questionnaire for the assessment of ICD-11 depression symptoms. Possible range of scores varies from 0 to 36. Higher scores indicate greater symptom severity.
Change in International Anxiety Questionnaire (IAQ) score | baseline; 10 weeks after randomization; 22 weeks after randomization; 32 weeks after randomization (delayed treatment group only)
  The IAQ is a self-report questionnaire for the assessment of ICD-11 anxiety symptoms. Possible range of scores varies from 0 to 32. Higher scores indicate greater symptom severity.
Change in World Health Organization Well-Being Index (WHO-5) score | baseline; 10 weeks after randomization; 22 weeks after randomization; 32 weeks after randomization (delayed treatment group only)
  The WHO-5 is a five-item self-report scale that assesses subjective psychological well-being. The range of the final WHO-5 index score ranges from 0 to 100, with higher scores indicating better well-being.
Change in Brief Version of the Posttraumatic Cognitions Inventory (PTCI-9) | baseline; 10 weeks after randomization; 22 weeks after randomization; 32 weeks after randomization (delayed treatment group only)
  PTCI-9 is a self-report measure assessing posttraumatic appraisals. The final score ranges from 9 to 63. Higher scale scores indicate stronger endorsement of negative cognitions.
Change in Trauma Related Shame Inventory - Short Form (TRSI-SF) | baseline; 10 weeks after randomization; 22 weeks after randomization; 32 weeks after randomization (delayed treatment group only)
  TRSI-SF is a self-report scale measuring trauma-related shame. The final score ranges from 0 to 30. Higher scores indicate higher levels of shame.
Patient satisfaction questionnaire (ZUF-8) | 10 weeks after randomization (immediate treatment group only); 32 weeks after randomization (delayed treatment group only)
  ZUF-8 is a self-report instrument for measuring patient satisfaction with the treatment/service received. The final score ranges from 8 to 32. Higher scores indicate stronger satisfaction with treatment.
Working Alliance Inventory for guided Internet Interventions (WAI-I) | 5 and 10 weeks after randomization (immediate treatment group only); 27 and 32 weeks after randomization (delayed treatment group only)
  WAI-I is a self-report instrument to assess the working alliance in the context of guided Internet interventions. The overall WAI-I score ranges from 12 to 60. Higher scores reflect stronger working alliance.
Readiness for Therapy Questionnaire (RTQ) | Baseline (before start using the intervention programme)
  RTQ is a self-report measure of clients' readiness for change. The final score ranges from 0 to 24. Higher scores indicate greater readiness for therapy.
The Treatment Expectation Questionnaire (TEX-Q) | Baseline (before start using the intervention programme)
  TEX-Q is a self-report assessment of clients' treatment expectations. The TEX-Q consists of 6 subscales: treatment benefit, positive impact, adverse events, negative impact, process, behavior control. Each item of the TEX-Q subscales is measured on a scale from 0 to 10. The mean score can range from 0 to 10. The overall score of TEX-Q is determined by calculating the mean with a reversal of the harm expectation subscales; higher values indicate more positive treatment expectations.

CONTACTS AND LOCATIONS:
Overall Officials: Odeta Gelezelyte, Dr., Principal Investigator — Vilnius University, Centre for Psychotraumatology

IPD SHARING:
Plan to Share IPD: Yes
Anonymized datasets used during the study will be available from the corresponding author upon reasonable request.
Supporting Information: Study Protocol
Time Frame: After the main results of the study are published.
Access Criteria: Anonymized datasets used during the study will be available from the corresponding author upon reasonable request.

REFERENCES:
- [Derived] Gelezelyte O, Guogaite G, Nomeikaite A, Bisson JI, Lewis C, Kazlauskas E. Efficacy of an internet-based guided trauma-focused intervention in reducing ICD-11 posttraumatic stress disorder symptoms: study protocol of a randomized controlled trial. BMC Psychiatry. 2024 Sep 30;24(1):645. doi: 10.1186/s12888-024-06097-0. PMID 39350097